CLINICAL TRIAL: NCT01369212
Title: Combination Therapy of Pegylated Interferon Alfa-2a and Tenofovir Versus Tenofovir Monotherapy in HBeAg-positive and HBeAg-negative Chronic Hepatitis B
Brief Title: Combination Therapy of Pegylated Interferon Alfa-2a and Tenofovir Versus Tenofovir Monotherapy in Chronic Hepatitis B
Acronym: HBRN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pittsburgh (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK082864 HBRN Immune Active; U01DK082864 (NIH); U01DK082843 (NIH); U01DK082863 (NIH); U01DK082866 (NIH); U01DK082867 (NIH); U01DK082871 (NIH); U01DK082872 (NIH); U01DK082874 (NIH); U01DK082919 (NIH); U01DK082923 (NIH); U01DK082927 (NIH); U01DK082943 (NIH); U01DK082944 (NIH); UL1TR000004 (NIH); UL1TR001111 (NIH); UL1TR000058 (NIH); P30DK050306 (NIH); A-DK-3002-001 (Other Grant/Funding Number: Interagency agreement with NIDDK); M01RR000040 (NIH); UL1RR024986 (NIH); NCT01821794 (obsolete NCT alias)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2022-10-12 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Hepatitis B Vaccines; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenofovir (Experimental): Tenofovir 192 weeks
  Interventions: Drug: Tenofovir
- Peginterferon-alfa 2a and tenofovir (Experimental): A combination of peginterferon-alfa 2a plus tenofovir for 24 weeks and then tenofovir only for 168 weeks
  Interventions: Drug: Peginterferon-alfa 2a and tenofovir

INTERVENTIONS:
Drug: Tenofovir — 300 mg daily for 192 weeks (4 years)
  Other Names: Hepatitis B; Viread
  Arms: Tenofovir
Drug: Peginterferon-alfa 2a and tenofovir — A combination of peginterferon-alfa 2a 180 µg weekly plus tenofovir 300 mg daily for 24 weeks and then only tenofovir 300 mg daily for 168 weeks (3.5 years).
  Other Names: Hepatitis B; PEGASYS; Viread; tenofovir
  Arms: Peginterferon-alfa 2a and tenofovir

SUMMARY:
This clinical trial compares the efficacy of peginterferon plus tenofovir for 24 weeks followed by monotherapy with tenofovir for a further 3.5 years to the efficacy of tenofovir alone given for 4 years in patients with chronic hepatitis B. The primary measure of outcome will be HBsAg loss in serum at 48 weeks after stopping all antiviral therapy (sustained off-treatment response).

DETAILED DESCRIPTION:
The objective of this study is to compare the long-term efficacy of treatment with combination therapy with peginterferon plus tenofovir versus tenofovir monotherapy in the treatment of chronic hepatitis B.

This is a randomized (1:1) parallel group design trial comparing (i) tenofovir disoproxil fumarate (TDF) 300 mg daily for 192 weeks (4 years) and (ii) peginterferon alfa-2a 180 µg weekly for 24 weeks plus Tenofovir DF 300 mg daily for 192 weeks (4 years). Enrolled participants will be stratified by HBeAg status (positive/negative), genotype (A vs. all others) and cirrhosis (present vs. absent). After 192 weeks of treatment, participants meeting criteria for treatment discontinuation will stop treatment and be followed for 48 weeks (total duration of treatment and follow up is 240 weeks). Emtricitabine/tenofovir coformulated as Truvada, approved for treatment of HIV but not for treatment of hepatitis B virus (HBV) infection, will be offered to patients with primary nonresponse, partial virological response or confirmed virologic breakthrough.

ELIGIBILITY:
Inclusion criteria:

* Participant is enrolled in the HBRN Cohort Study (NCT01263587) or completed the necessary components of the cohort baseline evaluation by the end of the baseline visit for this study
* 18 years or older
* Chronic hepatitis B infection as evidenced by at least one of the following:

  1. HBsAg positive result within 8 weeks prior to randomization and another time at least 24 weeks prior to randomization with no HBsAg negative result in between.
  2. HBsAg positive within 8 weeks prior to randomization and HBV DNA ≥1000 IU/mL on 2 occasions at least 24 weeks apart (can include result from screening visit within 8 weeks of randomization)
* Hepatitis B e antigen positive or negative
* Serum HBV DNA ≥1000 IU/mL on 2 occasions at least 4 weeks apart within the 32 weeks prior to randomization (can include result from screening visit within 8 weeks of randomization)
* At least 2 elevated serum alanine aminotransferase (ALT) levels (> 30 U/L for males, >20 U/L for females) 4 weeks apart, and no more than 32 weeks apart, with the second being within 8 weeks of randomization
* Compensated liver disease
* No evidence of hepatocellular carcinoma (HCC)
* Liver biopsy done that shows findings consistent with chronic hepatitis B with histology activity index (HAI) ≥3 (necroinflammatory component only) or Ishak fibrosis score ≥1 or both, as assessed by the local study pathologist on review of a liver biopsy done within 144 weeks of randomization
* Females of child bearing potential must agree to use an adequate method of contraception throughout the study and must have a negative pregnancy test immediately prior to the start of treatment

Exclusion criteria:

* Serum ALT ≥450 U/L for males and ≥300 U/L for females
* Treatment with interferon or nucleos(t)ide analogues for hepatitis B within 48 weeks of randomization
* More than 48 weeks of therapy with nucleos(t)ide analogues for hepatitis B at any time in the past
* History of hepatic decompensation including but not limited to ascites, variceal bleeding, or hepatic encephalopathy
* Known allergy or intolerance to any of the study medications
* Females who are pregnant or breastfeeding
* Previous organ transplantation including engrafted bone marrow transplant
* Any other concomitant liver disease, including hemochromatosis, hepatitis C or D; Participants with severe steatohepatitis will be excluded (participants with non-alcoholic fatty liver disease [NAFLD] with steatosis only and/or mild to moderate steatohepatitis are acceptable)
* Positive anti-HIV
* Renal insufficiency with calculated (by Modification of Diet in Renal Disease (MDRD) method) creatinine clearance <60 mL/min within 8 weeks prior to randomization
* Platelet count <90,000 /mm3, hemoglobin <13 g/dL (males) or <12 g/dL (females), absolute neutrophil count <1500 /mm^3 (<1000/mm^3 for African-Americans) within 8 weeks prior to randomization
* History of active alcohol or drug abuse within 48 weeks of screening.
* Pre-existing psychiatric condition(s), including but not limited to: Current moderate or severe depression as determined by the study physician, history of depression requiring hospitalization within past 10 years, history of suicidal or homicidal attempt within the past 10 years, or history of severe psychiatric disorders including but not limited to schizophrenia, psychosis, bipolar disorder
* History of immune-mediated disease, or cerebrovascular, chronic pulmonary or cardiac disease associated with functional limitation, retinopathy, uncontrolled thyroid disease, poorly controlled diabetes or uncontrolled seizure disorder
* Any medical condition that would be predicted to be exacerbated by therapy or that would limit study participation
* Any medical condition requiring or likely to require chronic systemic administration of corticosteroids or other immunosuppressive medications during the course of this study
* Evidence of active or suspected malignancy, or a history of malignancy within the last 144 weeks (except adequately treated carcinoma in situ or basal cell carcinoma of the skin)
* Need for ongoing use of any antivirals with activity against HBV during the course of the study
* Any other condition that in the opinion of the investigator would make the participant unsuitable for enrollment or could interfere with the participant participating in and completing the study.
* Participation in any other clinical trial involving investigational drugs within 30 days of randomization or intention to participate in another clinical trial during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-11; Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Averell Sherker, MD, Study Chair — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Edward Doo, MD, Study Chair — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Anna Lok, MD, Principal Investigator — University of Michigan
Locations (21):
- United States (20):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Queen's Medical Center, Honolulu, Hawaii
  - NIH Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- University of Toronto-Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository https://repository.niddk.nih.gov/home/
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- [Derived] Terrault NA, Sterling R, Lok AS, Ghany MG, Feld JJ, Cloherty G, Wahed AS, Yang X. Hepatitis B Virus RNA as a Biomarker for Safe Antiviral Discontinuation: A Prospective Study of Nucleos(t)ide Analogue Withdrawal. J Infect Dis. 2025 Jun 2;231(5):1290-1298. doi: 10.1093/infdis/jiae541. PMID 39478672
- [Derived] Feld JJ, Wahed AS, Fried M, Ghany MG, Di Bisceglie AM, Perrillo RP, Khalili M, Yang X, Belle SH, Janssen HLA, Terrault N, Lok AS; Hepatitis B Research Network (HBRN). Withdrawal of Long-Term Nucleotide Analog Therapy in Chronic Hepatitis B: Outcomes From the Withdrawal Phase of the HBRN Immune Active Treatment Trial. Am J Gastroenterol. 2023 Jul 1;118(7):1226-1236. doi: 10.14309/ajg.0000000000002176. Epub 2023 Jan 13. PMID 36728214
- [Derived] Terrault NA, Lok AS, Wahed AS, Ghany MG, Perrillo RP, Fried MW, Wong DK, Khalili M, Lau DTY, Sterling RK, Di Bisceglie AM, Lisker-Melman M, Cooper SL, Chung RT, Patel K, Roberts LR, Belle SH, Janssen HLA; Hepatitis B Research Network. Randomized Trial of Tenofovir With or Without Peginterferon Alfa Followed by Protocolized Treatment Withdrawal in Adults With Chronic Hepatitis B. Am J Gastroenterol. 2023 Jul 1;118(7):1214-1225. doi: 10.14309/ajg.0000000000002125. Epub 2022 Dec 23. PMID 36599136
- See also: Hepatitis B Research Network — http://www.hepbnet.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Started | 102 | 99
Completed | 95 | 92
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir | Total
Number analyzed (Participants) | 102 | 99 | 201
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41 [34 to 49] | 41 [34 to 50] | 41 [34 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 40 | 71
  Male | 71 | 59 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 80 | 85 | 165
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 9 | 7 | 16
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 21 | 22 | 43
  United States | 81 | 77 | 158
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Height data was missing for one participant
  kg/m^2
    number analyzed (Participants) | 101 | 99 | 200
    (all) | 25 [23 to 28] | 24 [22 to 27] | 24 [22 to 28]
HBeAg Positive [Count of Participants; unit: Participants] | 54 | 50 | 104
Quantitative HBeAg (qHBeAg) level [Median (Inter-Quartile Range); unit: log10 IU/mL] — Population: qHBeAg is measured only among HBeAg positive participants. One person in the Tenofovir group did not have this data
  log10 IU/mL
    number analyzed (Participants) | 54 | 49 | 103
    (all) | 3.0 [1.9 to 3.3] | 2.6 [1.6 to 3.2] | 2.9 [1.7 to 3.3]
Hepatitis B Virus (HBV) Genotype [Count of Participants; unit: Participants]
  A1 | 8 | 4 | 12
  A2 | 7 | 5 | 12
  B | 37 | 50 | 87
  C | 32 | 36 | 68
  D | 12 | 1 | 13
  E | 5 | 3 | 8
  F | 1 | 0 | 1
HBV DNA [Median (Inter-Quartile Range); unit: log10 IU/mL] | 6.7 [5.2 to 8.2] | 6.3 [5.2 to 7.9] | 6.5 [5.2 to 8.1]
Quantitative HBsAg level [Median (Inter-Quartile Range); unit: log10 IU/mL] | 3.9 [3.0 to 4.5] | 3.6 [3.0 to 4.9] | 3.8 [3.0 to 4.3]
ALT [Median (Inter-Quartile Range); unit: U/L] | 81 [56 to 133] | 71 [53 to 117] | 75 [55 to 119]
Platelet Count [Median (Inter-Quartile Range); unit: cells X 10^3/mm^3] | 192 [170 to 233] | 196 [161 to 227] | 193 [164 to 227]
Total Bilirubin [Median (Inter-Quartile Range); unit: mg/dL] | 0.6 [0.5 to 0.8] | 0.7 [0.5 to 0.8] | 0.6 [0.5 to 0.8]
White Cell Count [Median (Inter-Quartile Range); unit: cells X 10^3/mm^3] | 5.6 [4.8 to 6.5] | 5.2 [4.5 to 6.1] | 5.3 [4.5 to 6.2]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 14.8 [13.7 to 15.6] | 14.5 [13.7 to 15.6] | 14.6 [13.7 to 15.6]
Creatinine clearance [Median (Inter-Quartile Range); unit: mL/min/1.73m2] | 106 [93 to 117] | 96 [86 to 111] | 101 [90 to 117]
Albumin [Median (Inter-Quartile Range); unit: g/dL] — Population: One participant missing albumin levels
  g/dL
    number analyzed (Participants) | 101 | 99 | 200
    (all) | 4.2 [4.1 to 4.5] | 4.3 [4.0 to 4.6] | 4.3 [4.1 to 4.5]
Necroinflammatory Activity (HAI>= 3) [Count of Participants; unit: Participants] — Higher Ishak histological activity index (HAI) (necroinflammatory component only) indicates worse necroinflammatory activity [Possible range: 0 -18]. A score of 3 or higher indicates the presence of necroinflammatory activity.
  Participants | 97 | 96 | 193
Bridiging Fibrosis or Cirrhosis (Ishak score 5-6) [Count of Participants; unit: Participants] — Ishak fibrosis score (possible range 0-6) grades the fibrosis in the liver: 5 indicates bridging fibrosis and 6 indicates cirrhosis.
  Participants | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Hepatitis B Surface Antigen (HBsAg) Loss by Week 240
Description: Estimated percent of participants who became HBsAg negative by week 240 from randomization
Time Frame: Week 240
Population: This outcome is analyzed as a survival outcome with proportion estimated at week 240 using Kaplan-Meier Method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 102 | 99
Percentage of participants | 4.1 | 5.2
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.72, Wald test; Proportion with HBsAg loss at week 240 in each group is estimated by Kaplan-Meier and then equality of proportion is tested using Wald test

2. Secondary Outcome: Cumulative Percent of Participants With HBsAg Loss at Week 192
Description: Cumulative percentage of participants with HBsAg loss at week 192 estimated using Kaplan-Meier method
Time Frame: Week 192
Measure: Number; unit: Cumulative percentage of participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 102 | 99
Cumulative percentage of participants | 1.0 | 5.2
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.09, Wald Test — The cumulative percentages with HBsAg loss at week 192 were estimated using Kaplan-Meier method and then the equality is tested using Wald test

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with at least one serious adverse event between randomization and week 240
Time Frame: Up to 240 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 102 | 99
Participants | 11 | 7
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.46, Fisher Exact

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with at least one adverse event between randomization and week 240
Time Frame: up to 240 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 102 | 99
Participants | 50 | 60
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.12, Fisher Exact

5. Secondary Outcome: Number of Participants With Hepatitis B e Antigen (HBeAg) Loss at Week 192
Description: Number of participants who became Hepatitis B e antigen (HBeAg) negative at week 192 among HBeAg positive participants at randomization (baseline)
Time Frame: week 192
Population: Among HBeAg positive participants at baseline who had HBeAg data available at week 192
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 51 | 47
Participants | 14 | 29
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.002, Fisher Exact

6. Secondary Outcome: Number of Participants With HBeAg Loss at Week 240
Description: Number of participants who became HBeAg negative at week 240 among HBeAg positive participants at baseline
Time Frame: week 240
Population: Participants who were HBeAg positive at baseline and who had data for HBeAg at week 240 visit
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 49 | 45
Participants | 19 | 28
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.039, Fisher Exact

7. Secondary Outcome: Number of Participants With HBsAg Seroconversion at Week 192
Description: Number of participants who became with HBsAg negative and developed anti-HBs at week 192
Time Frame: week 192
Population: Participants with data on HBsAg and anti-HBs at week 192
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 96 | 92
Participants | 1 | 4
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.20, Fisher Exact

8. Secondary Outcome: Number of Participants With HBsAg Seroconversion at Week 240
Description: Number of participants who became HBsAg negative and developed anti-HBs at week 240
Time Frame: week 240
Population: HBsAg and antiHBs data at week 240
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 91 | 89
Participants | 2 | 4
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.44, Fisher Exact

9. Secondary Outcome: Number of Participants With HBeAg Seroconversion at Week 192
Description: Number of participants who became HBeAg negative and developed anti-HBe at week 192 among HBeAg positive participants at baseline
Time Frame: week 192
Population: HBeAg positives at baseline with HBeAg and anti-HBe data available at week 192
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 51 | 47
Participants | 8 | 16
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.06, Fisher Exact

10. Secondary Outcome: Number of Participants With HBeAg Seroconversion at Week 240
Description: Number of participants who became HBeAg negative and developed anti-HBe at week 240 among HBeAg positive participants at baseline
Time Frame: week 240
Population: HBeAg positive participants at baseline with HBeAg and anti-HBe data at week 240
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 49 | 45
Participants | 14 | 15
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.66, Fisher Exact

11. Secondary Outcome: Number of Participants With Normal Alanine Transaminase (ALT) Levels at Week 192
Description: Number of participants with normal alanine transaminase (ALT) levels at week 192 (Normal ALT for males ≤30 U/L, for females ≤20 U/L)
Time Frame: week 192
Population: Participants with ALT data at week 192
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 96 | 91
Participants | 37 | 51
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.02, Fisher Exact

12. Secondary Outcome: Number of Participants With Normal Alanine Transaminase (ALT) Levels at Week 240
Description: Number of participants with normal alanine transaminase (ALT) levels [males ≤30 U/L, for females ≤20 U/L] at week 240
Time Frame: week 240
Population: Participants with ALT data at week 240
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 92 | 89
Participants | 38 | 41
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.55, Fisher Exact

13. Secondary Outcome: Number of Participants With HBV DNA<1000 IU/mL at Week 192
Description: Number of participants with HBV DNA <1000 IU/mL at week 192
Time Frame: week 192
Population: Participants with HBV DNA data at week 192
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 96 | 91
Participants | 95 | 90
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p > 0.99, Fisher Exact

14. Secondary Outcome: Number of Participants With HBV DNA<1000 IU/mL at Week 240
Description: Number of participants with HBV DNA <1000 IU/mL at week 240
Time Frame: week 240
Population: Participants with HBV DNA data available at week 240
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 92 | 89
Participants | 66 | 65
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.87, Fisher Exact

15. Secondary Outcome: Number of Participants With HBV DNA<20 IU/mL at Week 192
Description: Number of participants with HBV DNA<20 IU/mL at week 192
Time Frame: week 192
Population: Participants with HBV DNA data at week 192
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 96 | 91
Participants | 82 | 87
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.02, Fisher Exact

16. Secondary Outcome: Number of Participants With HBV DNA<20 IU/mL at Week 240
Description: Number of participants with HBV DNA<20 IU/mL at week 240
Time Frame: week 240
Population: Participants with HBV DNA data at week 240
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 92 | 89
Participants | 46 | 48
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.66, Fisher Exact

17. Secondary Outcome: Absence of Detectable Antiviral Drug-Resistant HBV Mutations at Week 192
Description: Absence of detectable antiviral drug-resistant HBV mutations at Week 192
Time Frame: week 192
Population: The anti-viral drug resistance test was not done
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Cumulative Percent of Participants With HBsAg Loss at Week 240
Description: Cumulative percent of participants with HBsAg loss at week 240 estimated using Kaplan-Meier method
Time Frame: Week 240
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 102 | 99
percentage of participants | 4.1 | 5.2
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.66, Log Rank

19. Secondary Outcome: Number of Participants With Alanine Transaminase(ALT) Levels <= 38 U/L for Males and <=25 for Females at Week 192
Description: Number of participants with alanine transaminase(ALT) levels <= 38 U/L for males and <=25 for females at week 192. The cut-offs 38 and 25 are approximately 1.25 times the upper limit of normal (30 U/L for males and 20 U/L for females) respectively.
Time Frame: week 192
Population: Participants with ALT data at week 192
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
Number analyzed (Participants) | 96 | 91
Participants | 58 | 72
Statistical Analysis 1: Comparison: Tenofovir vs Peginterferon-alfa 2a and Tenofovir; Test type: Superiority; p = 0.01, Fisher Exact

ADVERSE EVENTS:
Time Frame: 240 weeks
Arm/Group | Tenofovir | Peginterferon-alfa 2a and Tenofovir
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/99
Serious Adverse Events (participants affected / at risk) | 11/102 | 7/99
Other Adverse Events (participants affected / at risk) | 50/102 | 60/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir (N=102) | Peginterferon-alfa 2a and Tenofovir (N=99)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
BENIGN PAROXYSMAL POSITIONAL VERTIGO (General disorders) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
CHEST PAIN (Cardiac disorders) | 1 (1) | 0 (0)
CHEST TIGHTNESS, LEFT SIDED WEAKNESS (Cardiac disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
CLINICAL DECOMPENSATION (Hepatobiliary disorders) | 1 (1) | 0 (0)
ELEVATED ALT (Hepatobiliary disorders) | 1 (1) | 0 (0)
FRACTURE, RIGHT ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GASTRECTOMY (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEARING LOSS (Nervous system disorders) | 0 (0) | 1 (2)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RECONSTRUCTION OF BREAST (Surgical and medical procedures) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
UTERINE FIBROIDS, OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir (N=102) | Peginterferon-alfa 2a and Tenofovir (N=99)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
BETA-THALESSEMIA, ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HYPOPHOSPHATEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
IRON DEFICIENCY DEVELOPED WITHOUT ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LOW ANC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LOW PLATELETS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LOW-NORMAL POTASSIUM LEVEL AND RUQ MUSCLE CRAMPS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
MICROCYTIC ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
PLATELET COUNT DECREASED (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
WHITE BLOOD CELL DECREASED (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
WHITE BLOOD CELL, PLATELET COUNT, AND NEUTROPHIL (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CHEST DISCOMFORT (Cardiac disorders) | 0 (0) | 1 (1)
CHEST PAIN (Cardiac disorders) | 0 (0) | 1 (1)
CHEST PRESSURE (Cardiac disorders) | 0 (0) | 1 (1)
HIGH CHOLESTEROL (Cardiac disorders) | 0 (0) | 1 (1)
HYPERTENSION (Cardiac disorders) | 2 (2) | 0 (0)
HYPERTENSION, DIZZINESS (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTRIGLYCERIDEMIA (Cardiac disorders) | 0 (0) | 1 (1)
RAPID HEART RATE (Cardiac disorders) | 0 (0) | 1 (1)
HEMOGLOBIN A1C ELEVATED (Endocrine disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
LOW TSH EPISODE (Endocrine disorders) | 0 (0) | 1 (1)
PARATHYROID ADENOMECTOMY (Endocrine disorders) | 1 (1) | 0 (0)
VITAMIN D DEFICIENCY (Endocrine disorders) | 1 (1) | 0 (0)
DRY EYES (Eye disorders) | 0 (0) | 1 (1)
PERIORBITAL EDEMA (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN, NAUSEA, GASTRIC REFLUX (Gastrointestinal disorders) | 0 (0) | 1 (1)
ACTIVE DUODENITIS WITH ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ACUTE APPENDICITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CAMPYLOBACTER INFECTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
CONSTIPATION, HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DAILY NAUSEA AND DIZZINESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DRY COUGH ASSOCIATED WITH EATING/REFLUX (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENDOSCOPIC ULTRASOUND SUGGESTED A SUBMUCOSAL GI TUMOR (GIST) (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIGASRIC PAIN AND BLACK DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS AND DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
H.PYLORI ANTIBODY POSITIVE (Gastrointestinal disorders) | 2 (2) | 0 (0)
HELICOBACTER PYLORI (Gastrointestinal disorders) | 0 (0) | 1 (1)
IRRITABLE BOWEL SYNDROME WITH DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA, MILD ABDOMINAL PAIN, WEAKNESS, DIZZINESS,SHORTNESS OF BREATH (Gastrointestinal disorders) | 1 (1) | 0 (0)
OPEN HERNIA UMBILICAL REPAIR (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPSET STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (1)
APHTHOUS ORAL ULCERS (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (1)
COUGH (General disorders) | 1 (1) | 1 (1)
DENTAL PROCEDURE (General disorders) | 1 (1) | 0 (0)
EAR ACHE POTENTIAL EAR INFECTION (General disorders) | 1 (1) | 0 (0)
EAR INFECTION/FUNGUS (General disorders) | 0 (0) | 1 (1)
EAR PAIN (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1)
FEVER (General disorders) | 1 (1) | 1 (1)
FLU-LIKE SYMPTOMS (General disorders) | 2 (3) | 2 (3)
HERPESVIRAL GINGIVOSTOMATITIS AND PHARYNGOTONSILLITIS (General disorders) | 0 (0) | 1 (1)
HYPOKALEMIA (General disorders) | 1 (1) | 0 (0)
INFECTION OF TOOTH (General disorders) | 2 (2) | 0 (0)
IRRITABILITY (General disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1)
MUCUS IN THROAT (General disorders) | 0 (0) | 1 (1)
NASAL CONGESTION AND POST NASAL DRIP (General disorders) | 0 (0) | 1 (1)
OTITIS EXTERNA (General disorders) | 0 (0) | 1 (1)
PREP (General disorders) | 1 (1) | 0 (0)
SINUSITIS (General disorders) | 0 (0) | 1 (1)
SURGICAL DENTAL EXTRACTION (General disorders) | 1 (1) | 0 (0)
TOOTH EXTRACTION (General disorders) | 0 (0) | 2 (2)
TOOTHACHE (General disorders) | 0 (0) | 1 (1)
ALT AND AST INCREASED (Hepatobiliary disorders) | 1 (1) | 1 (1)
ALT FLARE (Hepatobiliary disorders) | 3 (3) | 0 (0)
ELEVATED ALT (Hepatobiliary disorders) | 1 (1) | 3 (3)
ENLARGING GALLBLADDER POLYP (Hepatobiliary disorders) | 1 (1) | 0 (0)
HCC (Hepatobiliary disorders) | 1 (1) | 0 (0)
SEVERE FLARE DEVELOPED INTO CLINICAL DECOMPENSATION (Hepatobiliary disorders) | 1 (1) | 0 (0)
SPASM LIKE PAIN IN RUQ (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHEST PAIN (Immune system disorders) | 1 (1) | 0 (0)
RED ITCHY BUMPS/LESIONS ACROSS BODY (Immune system disorders) | 0 (0) | 1 (1)
SHINGLES (Immune system disorders) | 0 (0) | 1 (1)
SINUSITIS (Immune system disorders) | 1 (1) | 0 (0)
URTICARIA (Immune system disorders) | 0 (0) | 1 (1)
ACCIDENTAL OCCUPATIONAL BLOOD EXPOSURE TO HIV (Infections and infestations) | 1 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
SCRATCH BY CAT INFECTION AND PAIN (Infections and infestations) | 1 (1) | 0 (0)
SHINGLES (Infections and infestations) | 0 (0) | 1 (1)
SYPHILIS (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
WEIGHT LOSS (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
ACHES AND PAINS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ACUTE SCIATICA AND BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ANKLE FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (8) | 1 (1)
CERVICAL RADICULOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MOTORCYCLE ACCIDENT WITH MULTIPLE INJURIES (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — CONTUSION OF RIGHT SHOULDER AND HIP, SLAP TEAR OF GLENOID LABRUM, MINIMALLY DISPLACED RIGHT PUBIC ROOT W/NONDISPLACED INFERIOR PUBIC RAMUS FRACTURES AND SUSPECTED ANTERIOR LABRAL TEAR
ELBOW PAIN AND EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FOOT SPRAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GASTROCNEMIUS MUSCLE TEAR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INCREASED JOINT AND MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JOINT ACHES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
KNEE PAIN, LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LEFT KNEE EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PINCHED NERVE , NECK BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PROXIMAL HUMERUS FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RIGHT SHOULDER STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RIGHT TRIGGER AND MIDDLE FINGERS INCREASINGLY STIFF (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
THUMB PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TRIGGER MIDDLE FINGER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BELL'S PALSY (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
EPISODE OF SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 2 (2)
INSOMNIA (Nervous system disorders) | 0 (0) | 2 (2)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0)
NUMBNESS (Nervous system disorders) | 0 (0) | 1 (1)
ACUTE ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
DECREASED LIBIDO (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 6 (7)
HALLUCINATIONS (Psychiatric disorders) | 0 (0) | 1 (1)
INTERMITTENT CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 2 (2)
MOOD DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
MOOD SWING (Psychiatric disorders) | 0 (0) | 1 (1)
POLYNEUROPATHY (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL THOUGHT (Psychiatric disorders) | 0 (0) | 1 (1)
SYMPTOMS OF FEELING SAD, IRRITABLE, TROUBLE SLEEP (Psychiatric disorders) | 0 (0) | 1 (1)
BLOOD IN URINE (Renal and urinary disorders) | 1 (1) | 0 (0)
BPH WITH OBSTRUCTION/LOWER URINARY TRACT SYMPTOMS (Renal and urinary disorders) | 1 (1) | 0 (0)
DYSURIA, URINARY FREQUENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
E COLI INFECTION IN URINE (Renal and urinary disorders) | 1 (1) | 0 (0)
ERECTILE DYSFUNCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
KIDNEY STONE (Renal and urinary disorders) | 2 (2) | 1 (1)
LOW PHOSPHATE LEVELS (Renal and urinary disorders) | 1 (1) | 0 (0)
URETERIC STONE RECURRENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Renal and urinary disorders) | 3 (3) | 3 (3)
MENSES CEASED (Reproductive system and breast disorders) | 0 (0) | 1 (1) — PREGNANCY TESTS REMAINED NEGATIVE
POOR LIBIDO AND RECURRENT UTI (Reproductive system and breast disorders) | 0 (0) | 1 (1)
TUBAL REVERSAL (Reproductive system and breast disorders) | 0 (0) | 1 (1)
POST TUBAL REVERSION PROCEDURE WOUND INFECTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
MILD CHEST TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NON-PRODUCTIVE COUGH AND SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
REACTIVE AIRWAY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
CELLULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS HERPETIFORMIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DRY SKIN AND HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
EYE LID AND FACIAL SWELLING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HAIR LOSS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
HIVES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ITCHING (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
POISON IVY RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7)
RASH AT INJECTION SITE (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
RASH, SKIN IRRITATION, ERYTHEMA AT INJECTION SITE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
REDNESS AND ITCHINESS AT INJECTION SITE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RING WORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
TICK BITE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BACK SPRAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
From the Publications and Presentations policy "Disagreements between the HBRN Steering Committee and the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) on the merits of journal submission of a specific manuscript will be mediated through discussion on Steering Committee conference calls, ad hoc conference calls or during face to face Steering Committee meetings. The decision of the NIDDK is final and cannot be appealed."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT01369212/Prot_SAP_000.pdf